CLINICAL TRIAL: NCT02949674
Title: Ropivacaine Versus Bupivacaine as Preemptive Analgesia in Surgical Site in Ankle Fracture Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, JUAN LOPEZ VALENCIA, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-2016-3401-55
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2017-09

CONDITIONS: Ankle Fractures; Pain, Postoperative; Local Infiltration
MeSH Terms: conditions — Ankle Fractures; Pain, Postoperative | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Bupivacaine (Experimental): It will be used bupivacaine in surgical site prior surgery (25 mg). At least 10 minutes before skin incision.
  Interventions: Drug: Bupivacaine
- Ropivacaine (Experimental): It will be used ropivacaine in surgical site prior surgery (37.5 mg). At least 10 minutes before skin incision.
  Interventions: Drug: Ropivacaine
- Control (No Intervention): No application of anesthetic

INTERVENTIONS:
Drug: Ropivacaine — It will be used as a analgesic dose in surgical site before surgery.
  Other Names: Naropin
  Arms: Ropivacaine
Drug: Bupivacaine — It will be used as a analgesic dose in surgical site before surgery.
  Other Names: Bupivacaine hydrochloride
  Arms: Bupivacaine

SUMMARY:
Title: Ropivacaine versus Bupivacaine as Preventive Analgesia in Surgical Incision Site In Patients With Ankle Fracture Background: Ankle fractures are about 10% of the fractures associate to sports and with an incidence of 0.11 of 1000 adult patients. Weber classification system divides ankle fractures in three types according to the anatomy of lateral malleolus. B fractures starts at tibia pilon. Stable fractures are easily treated in conservative way. (12) Unstable fractures are treated surgically with anatomic reduction and internal fixation. However, it's been reported that even with successful reduction surgically great results are not always achieved. Local wound infiltration blocks the pain in its origin, surgical site by itself, without alter motor function. Practically without presenting adverse events with this method. it´s accurate for ambulatory surgery.

Main Objetive: To compare preventive analgesia with local anesthetic in surgical site with ropivacaine or bupivacaine in ankle fracture patients treated surgically with open reduction and internal fixation.

Method: Two groups with ankle fractures which will be informed and the patients will sign informed consent, after that the patients will be assign to a group (Ropivacaine or bupivacaine). The patient will be prepared for surgical treatment according to his doctor. It will be applied traditional anesthesia. It will be applied before beginning surgery in bupivacaine group 25 mg and in ropivacaine group 37.5 mg at least 10 minutes before starting surgery. After that the patient will have the traditional dose of analgesic treatment.The group will evaluate the pain with VAS 0-10 at 4,8,12 and 24 hours after surgery. The group will register data and will make statistic analysis. It will be elaborated the conclusion an elaboration of a report.

Resources: The group counts with human resources of the group of investigators. The hospital has in emergency department almost three patients with ankle fractures each day which require surgical treatment. The hospital has x ray service to valuate the ankle fracture and with computer system to analyze it. The hospital has the software for statistical analysis.

Experience: The group is formed with orthopedic surgeons with more than 5 years in treatment of ankle fractures. Investigators have the support of pain medicine group in hospital and with anesthesia coordinators. Investigators have a group of orthopedic residents which will be encharged of ilfiltration wound site.

Time: September 2016 to February 2017.

ELIGIBILITY:
Inclusion Criteria:

* Patient with afiliation to IMSS
* Patient with ankle fracture that requires surgical treatment with open reduction and internal fixation
* Patient that accept to participate in the study whit a sign of document.

Exclusion Criteria:

* Politrauma patients (Patients with another fracture)
* Patients who dont accept to participate in the study
* Neuropathy in inferior limps that limits pain perception
* Open ankle fractures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jonathan De La Cruz Pacheco, Study Chair — IMSS
Locations (1):
- UMAE Dr. Victorio de La Fuente Narvaez, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: January 2017 to April 2017, at High Specialty Unit Dr. Victorio de la Fuente Narvaez, IMSS
Period: Overall Study
Arm/Group | Bupivacaine | Ropivacaine | Control
Started | 31 | 31 | 31
Completed | 31 | 31 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Ropivacaine | Control | Total
Number analyzed (Participants) | 31 | 31 | 31 | 93
Age, Continuous [Mean (Full Range); unit: years] | 42.3 [18 to 67] | 37.16 [18 to 71] | 33.71 [18 to 67] | 37.7 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 17 | 51
  Male | 15 | 13 | 14 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 31 | 31 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: VAS
Description: The Pain will be measured with this scale from 0 (No pain) -10 (Worst pain possible) according to the investigator at 24 hours after surgery.
Time Frame: Change in Visual Analogue Scale at 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale (VAS)
Arm/Group | Bupivacaine | Ropivacaine | Control
Number analyzed (Participants) | 31 | 31 | 31
units on a scale (VAS)
  VAS at 4 hours | 2.81 (1.302) | 2.13 (0.619) | 3.52 (1.387)
  VAS at 8 hours | 4.52 (1.022) | 3.04 (1.113) | 5.02 (0.957)
  VAS at 12 hours | 4.42 (0.765) | 3.55 (0.995) | 4.84 (1.061)
  VAS at 24 hours | 4.03 (0.836) | 3.87 (0.783) | 4.10 (0.831)

ADVERSE EVENTS:
Arm/Group | Bupivacaine | Ropivacaine | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
We consider that we can had a better result with higher dosis of local anesthetic, and the comparation with a placebo group would be a better analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes